CLINICAL TRIAL: NCT02227472
Title: Working Memory and School Readiness in Preschool-Aged Children With Sickle Cell Disease: Family and Environmental Factors
Brief Title: Working Memory and School Readiness in Preschool-Aged Children With Sickle Cell Disease
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MEMREAD
Record Dates: First submitted 2014-08-22; First posted 2014-08-28 (Estimated); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sickle Cell Disease: All participants who meet eligibility requirements and consent to the study will complete evaluation of cognitive and pre-academic skills, and parent questionnaires.
  Interventions: Other: Evaluation of cognitive and pre-academic skills; Other: Parent questionnaires

INTERVENTIONS:
Other: Evaluation of cognitive and pre-academic skills — Participants will complete testing to evaluate fluid reasoning, knowledge, quantitative reasoning, visual-spatial processing, verbal and non-verbal working memory, and knowledge of pre-academic skills (such as colors, letters, numbers, counting, sizes, comparisons, and shapes).
  Other Names: Testing
Other: Parent questionnaires — Parents will complete questionnaires to assess behavioral manifestation of executive functions, functional independence and adaptive functioning, child and parent characteristics, situational/demographic life stress, demographics, education level, and household income.
  Other Names: Parent report

SUMMARY:
Children with sickle cell disease (SCD) are at risk for neurobehavioral problems because of the impact the disease can have on the central nervous system. Specific impairments in working memory are particularly prevalent in school-aged children with SCD. Working memory is more strongly associated with school readiness and academic success than intellectual ability in the general population. The adverse effects of low socioeconomic status (SES) and poverty on cognition and neurodevelopment emerge early, before children have entered formal education. In addition, they affect language and executive function skills (e.g., working memory) more than other skills. SES is a proxy variable for other risk factors. Higher SES is associated with less parental stress, more supportive parenting practices, and better cognitive stimulation based on the availability of books, computers, and outings.

PRIMARY OBJECTIVE:

* To examine working memory and school readiness in young children with sickle cell disease in comparison to demographically matched control children without sickle cell disease.

SECONDARY OBJECTIVE:

* To examine the relationships of family/environmental factors (caregiver stress, parental responsiveness, and cognitive stimulation in the home) and disease severity to working memory and school readiness skills in preschool-aged children with SCD.

DETAILED DESCRIPTION:
Participants will be recruited through the Pediatric Sickle Cell Clinic at St. Jude. All participants with SCD will be evaluated once with laboratory measures of cognitive and pre-academic skills and parent questionnaires. Medical history will be evaluated for purposes of characterizing the health status and disease severity of patients and determining how medical factors are related to school readiness and working memory in SCD population. The study expects to accrue up to 99 participants with SCD.

Demographically-matched control children will be selected from a database of participants enrolled in an ongoing longitudinal study of neurocognitive development in children born in Shelby County, Tennessee. The control group will be randomly selected from an existing study group and will not be enrolled on the MEMREAD protocol. Control group participants will be excluded if they have any sensory or motor impairment that would preclude valid testing (e.g., blindness, paresis), or if they have received treatment with non-stimulant psychotropic medication. A de-identified data file that includes the following results for up to 168 demographically-matched healthy control participants (approximately 1:2 ratio of SCD to healthy control) will be provided for control comparison purposes:

* Health Evaluation (CV4)
* Stanford binet - Fifth Edition (CV4)
* Bracken Basic Concepts Scale - Third Edition (CV4)
* The Behavior Rating Inventory of Executive Function - Preschool Version (BRIEF-P) (CV4)
* The Scales of Independent Behavior - Revised, Early Development Form (SIB-R) (CV4)
* Demographics (CV4)
* Additional Covariates (if any) including gestational age at birth, developmental delays, major medical illnesses, surgery history, neurological event history, pre-kindergarten attendance, and daycare attendance

ELIGIBILITY:
Inclusion Criteria:

* Patient at St. Jude Children's Research Hospital (SJCRH) with a primary diagnosis of sickle cell disease
* 48-68 months of age at time of enrollment
* English as primary language

Exclusion Criteria:

* Sensory or motor impairment that would preclude valid testing (e.g., blindness, paresis)
* Treatment with non-stimulant psychotropic medication
* Enrollment in kindergarten at time of assessment

Ages: 48 Months to 68 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants will be between 4 and 5 years of age, have a diagnosis of sickle cell disease (SCD) and be patients at St. Jude Children's Research Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2014-09-08 (Actual); Primary Completion 2018-08-20 (Actual); Study Completion 2018-08-20 (Actual)

PRIMARY OUTCOMES:
Mean difference in working memory between SCD participants and control group | Once, at enrollment
  Variables will be subjected to analyses to establish frequency distributions, means and standard deviations, and to determine if variables are normally distributed prior to use of parametric statistics. The primary dependent variable for working memory ability is the Working Memory Index from the SB-5. Primary dependent variables will be compared statistically using a paired sample one-side t-test.
Mean difference in school readiness between SCD group and control group | Once, at enrollment
  Variables will be subjected to analyses to establish frequency distributions, means and standard deviations, and to determine if variables are normally distributed prior to use of parametric statistics. The primary dependent variable for school readiness is the School Readiness Composite from the BBCS. Primary dependent variables will be compared statistically using a paired sample one-side t-test.
Association between working memory and school readiness skills compared between SCD group and control group | Once, at enrollment
  Variables will be subjected to analyses to establish frequency distributions, means and standard deviations, and to determine if variables are normally distributed prior to use of parametric statistics. Bivariate correlations will be used to investigate the association between working memory and school readiness skills.

SECONDARY OUTCOMES:
Effect of family/environmental factors and disease severity on measures of working memory | Once, within 6 months of enrollment
  Regression analyses will be used to examine the main effects of each family/environmental factor (caregiver stress, parental responsiveness, and cognitive stimulation in the home) and disease severity factors on measures of working memory and school readiness.
Effect of family/environmental factors and disease severity on school readiness | Once, within 6 months of enrollment
  Regression analyses will be used to examine the main effects of each family/environmental factor (caregiver stress, parental responsiveness, and cognitive stimulation in the home) and disease severity factors on measures of working memory and school readiness.

CONTACTS AND LOCATIONS:
Overall Officials: Jerlym Porter, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols